CLINICAL TRIAL: NCT06180434
Title: Short Term Outcomes After PRoton and PhotoN RadiOtherapy for IDH Mutated Grade 2 and 3 Gliomas
Acronym: SOPRANO
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Leiden University Medical Center (Other); HollandPTC (Industry); Institute Verbeeten (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Medical Center Groningen (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Maastro Clinic, The Netherlands (Other)
Responsible Party: Principal Investigator, Alejandra Mendez Romero, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2023-0727
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Glioma; Radiotherapy; Complications
Keywords: Neuro-oncology; Proton therapy; Photon therapy
MeSH Terms: conditions — Glioma | interventions — Proton Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Proton group: Patients with grade 2 and 3 IDHmt glioma treated with proton therapy in Holland PTC, Maastro Clinic and UMC Groningen.
  Interventions: Radiation: proton therapy
- Photon group: Patients with grade 2 and 3 IDHmt glioma treated with photon therapy in Erasmus MC, Haaglanden MC, LUMC, Amsterdam UMC locatie VUmc Site, Verbeeten Institute, Maastro Clinic, UMC Groningen, and Leuven University Hospital.
  Interventions: Radiation: photon therapy

INTERVENTIONS:
Radiation: proton therapy — Radiotherapy delivered with protons
  Groups: Proton group
Radiation: photon therapy — Radiotherapy delivered with photons
  Groups: Photon group

SUMMARY:
Rationale:

Proton beam therapy has recently become available for the treatment of patients with WHO grade 2 and 3 IDH mutated (IDHmt) glioma in the Netherlands. The dose distributions associated with proton therapy have substantially reduced the volume of the normal brain irradiated with low and intermediate radiotherapy doses. Whether this impacts rates of progressive disease or safety issues and how this compares with a similar population treated with photon therapy is currently unknown.

Objective:

To investigate short term outcomes after proton and photon radiotherapy for grade 2 and 3 IDHmt glioma.

DETAILED DESCRIPTION:
Patients with grade 2 and 3 IDHmt glioma treated with proton therapy in Holland PTC, Maastro and UMC Groningen and referred Erasmus MC, Haaglanden MC, LUMC, Amsterdam UMC, Verbeeten Institute, Maastro, UMC Groningen, and Leuven University Hospital between 1st of January 2018 and the 30th of June 2022. The outcomes will be compared to those from patients with grade 2 and 3 IDHmt glioma treated with photon therapy in the same institutes and during the same period of time. The applied clinical target volume (CTV) margins and the chemotherapy are preferably similar for proton and photon therapy.

Retrospective data will be collected from the electronic records of each participating institute. For the primary outcome, data will be collected on interventions (radiotherapy, surgery, chemotherapy, medication) for either tumor progression or toxicity after radiotherapy. This will be used to calculate next intervention free survival as primary outcome.

For the secondary outcomes, data on survival, disease progression, pseudoprogression, and toxicity will be used to calculate overall survival, progression free survival, and pseudoprogression free survival, as well as toxicity incidence.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed WHO grade 2 or grade WHO 3 IDHmt glioma
* Treatment with radiotherapy delivered between 1 of January 2018 and completed before or on the 30th of June 2022
* Treatment with chemotherapy delivered after radiotherapy (PCV or Temozolomide)
* Age ≥ 18 years

Exclusion Criteria:

* Prior cranial radiotherapy
* Contra-indication for MRI imaging
* Chemotherapy delivered before radiotherapy
* Dose and fractionation other that standard dose (50.4 Gy in 28 fractions for Grade 2 and 59.5 Gy in 33 fractions for Grade 3)
* Combination photon and proton therapy
* Patient has previously opted-out of the use of their data for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with proton radiation therapy for grade 2 and 3 IDHmt glioma referred to HollandPTC, Maastro and UMC Groningen from the 1st of January 2018 of and the 30th of June 2022. The photon group will consist of patients treated with photon radiation therapy within the same period in Erasmus MC, Haaglanden MC, LUMC, Amsterdam UMC, Verbeeten Institute, Maastro, UMC Groningen, and Leuven University Hospital. The reason for choosing this time interval is that the Dutch guideline for the treatment of glioma was updated regarding margins in December 2017. From January 2018 patients with grade 2 glioma were treated with a 5mm CTV margin to compensate for microscopic invasion. Patients with grade 3 IDHmt tumors were treated with 10mm CTV margins.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Next intervention-free survival | 24 months
  Time from the last day of radiotherapy until the start of a new next intervention. Next intervention is defined as either neurosurgical re-operation, re-irradiation, start of new chemotherapy (other than the standard adjuvant chemotherapy), start of VGEF inhibitors such as bevacizumab, or new start of dexamethasone for either tumor progression or radiotherapy effects.

SECONDARY OUTCOMES:
Adverse Events | 24 months
  Assessed and scored based on the Common Terminology Criteria for Adverse Events (CTCAEv5.0). Only grade 3, 4 and 5 adverse events will be recorded.
Overall survival | 24 months
  Measured from the last day of radiotherapy to death from any cause
Progression-free survival | 24 months
  Time from the last day of radiotherapy until progressive disease
Pseudoprogression-free survival | 24 months
  time from the last day of radiotherapy and the development of any transient contrast-enhancing lesion between the end of radiotherapy and disease progression, or any new contrast-enhancing lesion that remained stable over a period of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Mendez Romero, MD PhD, Principal Investigator — Assitant Professor, Radiation Oncologist
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No